CLINICAL TRIAL: NCT03433144
Title: The Effects of Tranexamic Acid on Blood Loss During Orthognathic Surgery
Acronym: TXA-OMFS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Nick Emanuele (Other)
Responsible Party: Sponsor-Investigator, Nick Emanuele, Resident, Oral and Maxillofacial Surgery, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1023246
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Tranexamic Acid; Orthognathic Surgery

STUDY DESIGN:
Intervention Model Description: In this study, patients will be randomized into two groups: and intervention group and placebo. The intervention group will receive a single pre-operative dose of TXA IV (10mg/kg) and the placebo group will receive the same volume of fluid intravenously.
Who Masked: Participant
Masking Description: The patient will be unaware of which group they have been randomized into
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention TXA (Experimental): patients receiving TXA10mg/kg IV pre-operatively
  Interventions: Drug: Tranexamic Acid Injectable Solution
- Placebo (Placebo Comparator): patients will receive an equivalent amount of normal saline 0.9% IV pre-operatively
  Interventions: Other: Placebo (normal saline 0.9%)

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Solution — the drug will be given to patients intravenously at a dose of 10mg/kg pre-operatively after induction on general anesthesia
  Arms: Intervention TXA
Other: Placebo (normal saline 0.9%) — An equivalent amount of normal saline (0.9%) will be given to the patient pre-operatively after induction of general anesthesia. The amount of saline given will correspond to the same amount of fluid which would have been given had the patient been in the intervention group.
  Arms: Placebo

SUMMARY:
This study seeks to answer the question: Does a single pre-operative dose of tranexamic acid have a statistically significant reduction in blood loss during orthognathic surgery?

If it does, this drug may begin to be used routinely during orthognathic surgery to reduce blood loss in our patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing either

  * Bilateral saggital split osteotomy (lower jaw surgery)
  * Lefort 1 osteotomy (upper jaw surgery)
  * Combination of BSSO and Lefort
* Patients between with ages of 16-65
* No cardiac comorbidities (hypertension, congenital heart malformation)
* No known coagulopathy
* No regular prescription medication altering normal blood coagulation (NSAIDs, other anticoagulants)
* ASA I and II patients

Exclusion Criteria:

* Patients younger than 16 and older than 40
* Patients with known coagulopathy
* Patients with cardiac comorbidities
* Patients with a family history of bleeding disorders
* Patients who have undergone previous orthognathic surgery
* ASA III patients or higher

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
blood loss during surgery | intra-operative only
  meticulous measurement of the total blood loss encountered during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nick Emanuele, DDS, BBA, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
The data will be used for internal use only